CLINICAL TRIAL: NCT02983526
Title: Randomized Controlled Study Comparing a Short Stem Hip Prosthesis With a Stem of Standard Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johan Karrholm (Other)
Responsible Party: Sponsor-Investigator, Johan Karrholm, MD, Professor in Orthopaedics, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFP-SUH
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Primary Osteoarthritis of Hip Nos; Secondary Osteoarthritis of Hip
Keywords: short stem
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Total hip replacement (2 different designs) — Patients will randomly receive either CFP or Corail stem
  Other Names: CFP stem or Corail stem

SUMMARY:
80 patients eligible for a total hip replacement (THR) mainly due to primary osteoarthritis were recruited from the waiting list for hip arthroplasty at a university hospital in Sweden. The patients were randomized to either CFP or Corail stem, both groups received Delta cup from Lima. Randomisation was done using envelopes. Patients could only participate with one hip. Patients are evaluated with different questionnaires, radiographs and RSA analysis.

DETAILED DESCRIPTION:
The concept of femoral neck preserving hip replacement is intended for the young and active patients. By preserving proximal bone load, the transmission to the proximal femur is supposed to improve and future revision surgery would be facilitated. The hypothesis is that a more conservative resection of the femoral neck could lead to better clinical outcomes compared to a conventional stem. The clinical outcomes and the fixation of a short femoral stem were therefore compared with a stem of standard length. 83 patients were included in our randomized controlled trial where patients either received a Collum Femoris Preserving (CFP) stem or a Corail hip stem. Clinical outcomes are being assessed, plain radiographs are studied and the early migration is being measured using radiostereometric analysis. All of the patients have gone through 1 year follow-up. The 2 years results will be available at the end of 2017.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis of hip
* secondary osteoarthritis due to hip dysplasia or Perthes under condition that the collum anatomy is well preserved and largely unaffected by the primary disease
* avascular necrosis of femoral head
* anatomy suitable for both designs according to preoperative planning

Exclusion Criteria:

* previous treatment with cortisone
* generalized joint disease

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Oxford Hip Score | Preoperatively to 2 years
  The Oxford Hip Score (OHS) is a short 12-item patient-reported PRO specifically designed and developed to assess function and pain with patients undergoing hip replacement surgery. It is short, reproducible, valid and sensitive to clinically important changes.
Radiostereometric analysis | Preoperatively to 2 years
  Radiostereometric analysis is an accurate method of determining the migration and wear of orthopaedic implants such as total hip arthroplasties. The overall concept of RSA is straightforward: determining the precise location of two distinct objects relative to each other in three dimension (such as the relative position of the femoral component and the proximal femur).

SECONDARY OUTCOMES:
Patient satisfaction (VAS), Pain (VAS) | Preoperatively to 2 years
  Patient satisfaction and pain are reported on visual analogue scales.
Harris hip score | Preoperatively to 2 years
  One of the oldest and most commonly used scores to assess function and pain with patients undergoing hip replacement surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Kärrholm, MD, PhD, Professor, Principal Investigator — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: Undecided